CLINICAL TRIAL: NCT04724408
Title: Endotracheal Intubation With VieScope Versus Direct Laryngoscopic Intubation in Patients for Elective Surgery - a Prospective Randomized Trial.
Brief Title: VieScope Versus Direct Laryngoscopic Intubation
Acronym: VieScOP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VieScOP
Record Dates: First submitted 2021-01-23; First posted 2021-01-26 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Airway Management

STUDY DESIGN:
Intervention Model Description: randomized 1:1
Who Masked: Participant
Masking Description: device for intubation may not be blinded for provider or investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VieScope (Experimental): intubation with the VieScope laryngoscope
  Interventions: Device: VieScope
- Conventional (Active Comparator): intubation with MacIntosh-type laryngoscope
  Interventions: Device: Conventional

INTERVENTIONS:
Device: VieScope — see above
  Arms: VieScope
Device: Conventional — see above
  Arms: Conventional

SUMMARY:
Patients requiring endotracheal intubation for elective surgery without expected difficult airway are randomized to be intubated either by a) VieScope or b) conventional direct laryngoscopy.

DETAILED DESCRIPTION:
Endotracheal intubation is required for different surgical procedures for mechanical ventilation and to prevent aspiration of secretions. Endotracheal intubation is usually performed by direct laryngoscopy (DL), i.e. during otorhinolaryngologic or oral and maxillofacial surgery. This technique has limitations and may fail due to insufficient visualization of the larynx. A new device has been introduced that consists of an illuminated straight plastic tube for laryngoscopy (VSC, Vie Scope, Adroit Surgical, Oklahoma City, OK, USA) that enables for indirect intubation over a stylet. So far, the VSC has shown promising results in manikin studies for intubation in normal and difficult airways and was shown to be superior over conventional laryngoscopy during cardiopulmonary resuscitation with providers wearing personal protective equipment. Data in elective patients undergoing otorhinolaryngologic or oral and maxillofacial surgery are not available, so far.

Therefore, we aim to test the VSC in patients compared to conventional techniques in a prospective randomized non-inferiority trial. We aim to test the VSC in predicted non-difficult airway patients.

Patients will be assessed for eligibility in the Anesthesiology Pre-assessment Clinic of the University Medical Center Hamburg-Eppendorf prior to elective surgery. To rule out a difficult airway prior to study inclusion, all patients receive a structured preoperative airway assessment in accordance with standard operating procedure of the Department of Anesthesiology, University Medical Center Hamburg-Eppendorf using the implemented in-house algorithm for the prediction of difficult airway management and the Simplified Airway Risk Index (SARI).

Patients are randomized 1:1 to either intervention or control group. Patients randomized to the intervention group will be intubated with the VSC. Patients randomized to the control group are intubated with a standard MacIntosh type laryngoscope by DL. Anesthesia management, the choice of the blade and tube size, as well as the use of adjuncts like stylets, introducers or forceps or airway optimization maneuvers (e.g. backward upward rightward pressure [BURP] and optimum external laryngeal manipulation [OELM]) will be left to the discretion of the attending physician.

Based on a first attempt success rate of 40%, and a noninferiority margin of 5%, 2x 29 patients are required with errors of α=0.025 and β=0.2 to show non-inferiority for the intervention method (PASS version 08.0.6, NCSS, LLC. Kaysville, UT, USA).

All participating physicians are anesthesiology residents or fellows. To avoid a bias that may occur due to different skills for VSC compared to conventional laryngoscopy, physicians participating in this study take part in a 30 min structured manikin airway training before participating in this study. The age and months of work experience of the participating anesthetists will be assessed within a questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring general anesthesia with transoral tracheal intubation for elective surgery
* Age ≥ 18
* Preoperative airway assessment reveals an expected non-difficult airway (rated by the responsible anesthetist in the Pre-assessment Clinic based on the existing in-house algorithm)

Exclusion Criteria:

* Pregnant or breastfeeding woman
* Confirmed indications for awake fiberoptic intubation especially due to enoral, pharyngeal tumors, abscesses or other processes
* Planned endotracheal intubation without deep anesthesia or neuromuscular blocking agents (e.g. awake videolaryngoscopy)
* Required transnasal tracheal intubation (e.g. for surgical reasons)
* Requirement of special endotracheal tubes such as laser or RAE tubes for surgical reasons
* Patients at risk for pulmonary aspiration who qualify for rapid sequence induction
* Loose teeth
* Denial of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2021-01-26 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
First attempt success rate | 15 min
  percentage of successful intubations with one attempt

SECONDARY OUTCOMES:
intubating conditions | 15 min
  grades according to Cormack-Lehane and POGO
overall success rate | 15 min
  percentage of successful intubations with the allocated procedure
time to successful intubation | 15 min
  time until an endotracheal airway access is established
time to successful intubation with one attempt | 15 min
  time until an endotracheal airway access is established in patients that are intubated at first attempt
intubation difficulty | 15 min
  subjective rating on a visual analogue scale (0-100, higher values indicate more difficult intubation) of the difficulty of airway management and questionnaire
end-tidal carbondioxide fraction | 15 min
  the highest end-tidal carbondioxide fraction in the exspiratory gas within two minutes after successful intubation
number of attempts | 15 min
  total number of attempts until airway established
aspiration | 15 min
  percentage of patients that vomit and aspirate during intubation
esophageal intubation | 15 min
  percentage of accidental esophageal intubation attempts
hypoxia | 15 min
  percentage of patients with a desaturation below a pulsoximetric saturation of 80%
hypotension | 15 min
  percentage of patients with a systolic blood pressure below 70 mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Joern Grensemann, MD, Study Chair — Universitätsklinikum Hamburg-Eppendorf; Martin Petzoldt, MD, Study Chair — Universitätsklinikum Hamburg-Eppendorf
Locations (1):
- Universitätsklinikum Hamburg-Eppendorf, Hamburg, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: Undecided